CLINICAL TRIAL: NCT03859518
Title: Study of the Role of Innate Lymphoid Cells and Natural Killer Cells in Immune Activation of Vitiligo
Brief Title: Study of the Role of Innate Lymphoid Cells and Natural Killer Cells in Immune Activation of Vitiligo - INNATE Vitiligo
Acronym: INNATEvitiligo
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 18-GIRCI-01
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-01

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with Vitiligo
  Interventions: Other: blood and skin samples
- control
  Interventions: Other: blood and skin samples

INTERVENTIONS:
Other: blood and skin samples — To study the presence and type of ILC and NK in the blood and skin of vitiligo patients compared to control subjects.

SUMMARY:
The cohort included only major patients with non-segmental vitiligo and no other autoimmune or inflammatory associated diseases (except thyroiditis). Control subjects should have no autoimmune or inflammatory diseases. Patients and controls should not take treatment with corticosteroids or other potentially immunomodulatory therapies. Patients and controls are recruited in the Dermatology Department of the University Hospital of Nice and the Hospital of Fréjus. The investigators have already initiated the collection of tissues and blood from patients and control subjects and we have succeeded in isolating ILCs and NKs from a blood volume of 50ml. We were able to sort the ILC subpopulations. Early data suggest an increase in Natural Killer (NK) and Innate Lymphoïdes Cells 1 (ILC1) in the blood of vitiligo patients compared to control subjects. The investigators also managed to extract the melanocytes from the skin biopsies of the first patients and control subjects.

DETAILED DESCRIPTION:
The investigators want study the presence and type of ILC and NK in the blood and skin of vitiligo patients compared to control subjects.

ELIGIBILITY:
Inclusion Criteria:

vitiligo subjects :

* patients in the cohort with non-segmental vitiligo
* without other autoimmune or inflammatory diseases associated

control subjects :

* subject without autoimmune or inflammatory disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: in this study, there are 2 groups. First with vitiligo and the second only with control subjects without autoimmune or inflammatory diseases.
  All this subjects were include in the dermatolgy servive of the CHU of Nice.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
study the presence and type of ILC and NK in the blood and skin | 1 day
  Compare vitiligo patients to control subjects.
study the presence and type of ILC and NK in the skin | 1 day
  Compare vitiligo patients to control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PASSERON, MD; PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CH de Frejus, Fréjus, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spritz RA. Six decades of vitiligo genetics: genome-wide studies provide insights into autoimmune pathogenesis. J Invest Dermatol. 2012 Feb;132(2):268-73. doi: 10.1038/jid.2011.321. Epub 2011 Oct 13. PMID 21993561
- [Background] Jin Y, Birlea SA, Fain PR, Ferrara TM, Ben S, Riccardi SL, Cole JB, Gowan K, Holland PJ, Bennett DC, Luiten RM, Wolkerstorfer A, van der Veen JP, Hartmann A, Eichner S, Schuler G, van Geel N, Lambert J, Kemp EH, Gawkrodger DJ, Weetman AP, Taieb A, Jouary T, Ezzedine K, Wallace MR, McCormack WT, Picardo M, Leone G, Overbeck A, Silverberg NB, Spritz RA. Genome-wide association analyses identify 13 new susceptibility loci for generalized vitiligo. Nat Genet. 2012 May 6;44(6):676-80. doi: 10.1038/ng.2272. PMID 22561518
- [Background] Jin Y, Andersen G, Yorgov D, Ferrara TM, Ben S, Brownson KM, Holland PJ, Birlea SA, Siebert J, Hartmann A, Lienert A, van Geel N, Lambert J, Luiten RM, Wolkerstorfer A, Wietze van der Veen JP, Bennett DC, Taieb A, Ezzedine K, Kemp EH, Gawkrodger DJ, Weetman AP, Koks S, Prans E, Kingo K, Karelson M, Wallace MR, McCormack WT, Overbeck A, Moretti S, Colucci R, Picardo M, Silverberg NB, Olsson M, Valle Y, Korobko I, Bohm M, Lim HW, Hamzavi I, Zhou L, Mi QS, Fain PR, Santorico SA, Spritz RA. Genome-wide association studies of autoimmune vitiligo identify 23 new risk loci and highlight key pathways and regulatory variants. Nat Genet. 2016 Nov;48(11):1418-1424. doi: 10.1038/ng.3680. Epub 2016 Oct 10. PMID 27723757
- [Background] Chatterjee S, Eby JM, Al-Khami AA, Soloshchenko M, Kang HK, Kaur N, Naga OS, Murali A, Nishimura MI, Caroline Le Poole I, Mehrotra S. A quantitative increase in regulatory T cells controls development of vitiligo. J Invest Dermatol. 2014 May;134(5):1285-1294. doi: 10.1038/jid.2013.540. Epub 2013 Dec 23. PMID 24366614
- [Background] Mosenson JA, Zloza A, Nieland JD, Garrett-Mayer E, Eby JM, Huelsmann EJ, Kumar P, Denman CJ, Lacek AT, Kohlhapp FJ, Alamiri A, Hughes T, Bines SD, Kaufman HL, Overbeck A, Mehrotra S, Hernandez C, Nishimura MI, Guevara-Patino JA, Le Poole IC. Mutant HSP70 reverses autoimmune depigmentation in vitiligo. Sci Transl Med. 2013 Feb 27;5(174):174ra28. doi: 10.1126/scitranslmed.3005127. PMID 23447019
- [Background] Harris JE, Harris TH, Weninger W, Wherry EJ, Hunter CA, Turka LA. A mouse model of vitiligo with focused epidermal depigmentation requires IFN-gamma for autoreactive CD8(+) T-cell accumulation in the skin. J Invest Dermatol. 2012 Jul;132(7):1869-76. doi: 10.1038/jid.2011.463. Epub 2012 Feb 2. PMID 22297636
- [Background] Rashighi M, Agarwal P, Richmond JM, Harris TH, Dresser K, Su MW, Zhou Y, Deng A, Hunter CA, Luster AD, Harris JE. CXCL10 is critical for the progression and maintenance of depigmentation in a mouse model of vitiligo. Sci Transl Med. 2014 Feb 12;6(223):223ra23. doi: 10.1126/scitranslmed.3007811. PMID 24523323
- [Background] Boniface K, Jacquemin C, Darrigade AS, Dessarthe B, Martins C, Boukhedouni N, Vernisse C, Grasseau A, Thiolat D, Rambert J, Lucchese F, Bertolotti A, Ezzedine K, Taieb A, Seneschal J. Vitiligo Skin Is Imprinted with Resident Memory CD8 T Cells Expressing CXCR3. J Invest Dermatol. 2018 Feb;138(2):355-364. doi: 10.1016/j.jid.2017.08.038. Epub 2017 Sep 18. PMID 28927891
- [Background] Yu R, Broady R, Huang Y, Wang Y, Yu J, Gao M, Levings M, Wei S, Zhang S, Xu A, Su M, Dutz J, Zhang X, Zhou Y. Transcriptome analysis reveals markers of aberrantly activated innate immunity in vitiligo lesional and non-lesional skin. PLoS One. 2012;7(12):e51040. doi: 10.1371/journal.pone.0051040. Epub 2012 Dec 10. PMID 23251420
- [Background] Regazzetti C, Joly F, Marty C, Rivier M, Mehul B, Reiniche P, Mounier C, Rival Y, Piwnica D, Cavalie M, Chignon-Sicard B, Ballotti R, Voegel J, Passeron T. Transcriptional Analysis of Vitiligo Skin Reveals the Alteration of WNT Pathway: A Promising Target for Repigmenting Vitiligo Patients. J Invest Dermatol. 2015 Dec;135(12):3105-3114. doi: 10.1038/jid.2015.335. Epub 2015 Aug 31. PMID 26322948
- [Background] Bernardini G, Gismondi A, Santoni A. Chemokines and NK cells: regulators of development, trafficking and functions. Immunol Lett. 2012 Jul 30;145(1-2):39-46. doi: 10.1016/j.imlet.2012.04.014. PMID 22698182
- [Background] Bruggen MC, Bauer WM, Reininger B, Clim E, Captarencu C, Steiner GE, Brunner PM, Meier B, French LE, Stingl G. In Situ Mapping of Innate Lymphoid Cells in Human Skin: Evidence for Remarkable Differences between Normal and Inflamed Skin. J Invest Dermatol. 2016 Dec;136(12):2396-2405. doi: 10.1016/j.jid.2016.07.017. Epub 2016 Jul 22. PMID 27456756